CLINICAL TRIAL: NCT01792817
Title: Non-invasive Neurostimulation of the Vagus Nerve With the GammaCore Device for the Treatment of Cluster Headache
Brief Title: Non-invasive Neurostimulation of the Vagus Nerve for the Treatment of Cluster Headache
Acronym: CH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ElectroCore INC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CH-US-01
Record Dates: First submitted 2013-02-08; First posted 2013-02-15 (Estimated); Results first posted 2018-05-17 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Cluster Headache
Keywords: Cluster Headache; GammaCore; vagal nerve stimulation; nVNS; VNS; non invasive; vagus nerve stimulation
MeSH Terms: conditions — Cluster Headache

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sham GammaCore device (Sham Comparator): The Sham GammaCore device looks and operates like the Active GammaCore device, but does not deliver a therapeutic stimulation treatment.
  Interventions: Device: Sham GammaCore device
- GammaCore Device (Experimental): Non-Invasive Vagus Nerve Stimulator
  Interventions: Device: GammaCore

INTERVENTIONS:
Device: GammaCore — Treatment with active gammacore vagus nerve stimulator
  Arms: GammaCore Device
Device: Sham GammaCore device — Treatment with sham stimulator
  Arms: Sham GammaCore device

SUMMARY:
Multi-center, prospective, double-blind, randomized, sham-controlled pivotal study of non-invasive vagus nerve stimulation with the GammaCore® device for the acute treatment of cluster headache. The study compares the safety and effectiveness of an active treatment (GammaCore) against a sham treatment.

DETAILED DESCRIPTION:
Phase 1: Prospective, randomized (1:1 active treatment:sham control allocation), double blinded, sham controlled treatment (active or sham) phase

Phase 2: Prospective, non-randomized, active treatment phase.

Phase 1 - Two Arms:

1. Active Treatment with the GammaCore Device
2. Sham Treatment with a placebo device

Phase 2 - One Arm:

Active Treatment with the GammaCore Device

ELIGIBILITY:
Inclusion Criteria:

1. Is between the ages of 18 and 75 years.
2. Has been diagnosed with cluster headache, in accordance with the ICHD-2

   Classification criteria (2ndEd):

   o At least 5 attacks fulfilling the following criteria:
   * Severe or very severe unilateral orbital, supraorbital and/or temporal pain lasting 15-180 minutes if untreated
   * Headache is accompanied by at least 1 of the following:
   * Ipsilateral conjunctival injection and/or lacrimation
   * Ipsilateral nasal congestion and/or rhinorrhea
   * Ipsilateral eyelid edema
   * Ipsilateral forehead and facial sweating
   * Ipsilateral miosis and/or ptosis
   * A sense of restlessness or agitation
3. currently experiencing cluster headaches, and from clinical history is expected to continue experiencing cluster headaches for a period of at least 4 weeks.
4. able to distinguish CH from other headaches (i.e. migraine, tension-type headaches).
5. capable of completing headache pain self-assessments.
6. [Intentionally left blank].
7. Agrees to use the GammaCore device as intended and follow all of the requirements of the study, including follow-up visit requirements.
8. Agrees to record usage of the GammaCore device, all required study data, and report any adverse device effects to the study center within 24 hours of any such adverse device effects.
9. able to provide written Informed Consent

Exclusion Criteria:

1. had surgery to treat cluster headache.
2. currently taking prophylactic medication (including chronic opioids and non-prescribed street drugs) for indications other than CH that in the opinion of the clinician may interfere with the study.
3. [Intentionally left blank].
4. undergone botulinum toxin injections in the head and/or neck in the last 3 months or nerve blocks (occipital or other) in the head or neck in the last month.
5. history of aneurysm, intracranial hemorrhage, brain tumors or significant head trauma.
6. lesion (including lymphadenopathy), dysaesthesia, previous surgery or abnormal anatomy at the treatment site.
7. structural intracranial, or cervical vascular lesions that may potentially cause headache attacks.
8. other significant pain problem (including cancer pain, fibromyalgia, and trigeminal neuralgia/TAC-cluster) that might confound the study assessments.
9. known or suspected severe atherosclerotic cardiovascular disease, severe carotid artery disease (e.g. bruits or history of TIA or CVA), congestive heart failure (CHF), known severe coronary artery disease or recent myocardial infarction.
10. history of prolonged QT interval or a history of clinically significant arrhythmia.
11. abnormal baseline ECG (e.g. second and third degree heart block, atrial fibrillation, atrial flutter, recent history of ventricular tachycardia or ventricular fibrillation, or clinically significant premature ventricular contraction).
12. previous bilateral or right cervical vagotomy.
13. uncontrolled high blood pressure.
14. currently implanted with an electrical and/or neurostimulator device, including but not limited to cardiac pacemaker or defibrillator, vagal neurostimulator, deep brain stimulator, spinal stimulator, bone growth stimulator, or cochlear implant.
15. history of carotid endarterectomy or vascular neck surgery on the right side.
16. implanted with metal cervical spine hardware or has a metallic implant near the GammaCore stimulation site.
17. recent or repeated history of syncope.
18. recent or repeated history of seizure.
19. known history or suspicion of substance abuse or addiction, or overuse of acute headache medication for headaches other than CH.
20. psychiatric or cognitive disorder and/or behavioral problems which in the opinion of the clinician may interfere with the study.
21. pregnant, nursing, thinking of becoming pregnant in the next 4 months, or of childbearing years and is unwilling to use an accepted form of birth control.
22. participating in any other therapeutic clinical investigation or has participated in a clinical trial in the preceding 30 days.
23. Belongs to a vulnerable population or has any condition such that his or her ability to provide informed consent, comply with follow-up requirements, or provide self-assessments is compromised

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2013-02; Primary Completion 2014-06 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lia Spitzer, Study Director — ElectroCore INC
Locations (20):
- United States (20):
  - California Medical Clinic for Headache, Santa Monica, California
  - Stanford University Medical Center, Stanford, California
  - Colorado Neurological Institute, Englewood, Colorado
  - Associated Neurologists of Southern Connecticut, Fairfield, Connecticut
  - Tampa General Hospital Headache Center, Tampa, Florida
  - Diamond Headache Clinic, Chicago, Illinois
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - Norton Neurology, Louisville, Kentucky
  - Mid-Atlantic Headache Institute, Pikesville, Maryland
  - New England Regional Headache Center, Worcester, Massachusetts
  - Michigan Head Pain & Neurological Institute, Ann Arbor, Michigan
  - Headache Care Center, Springfield, Missouri
  - Dent Neurologic Institute, Amherst, New York
  - Montefiore Headache Center, New York, New York
  - Center for Headache Care and Research at Island Neurological Associates, PC, Plainview, New York
  - Carolina Headache Institute, Chapel Hill, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Jefferson Headache Center, Philadelphia, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
  - West Virginia University Dept of Neurology, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Coo IF, Marin JC, Silberstein SD, Friedman DI, Gaul C, McClure CK, Tyagi A, Liebler E, Tepper SJ, Ferrari MD, Goadsby PJ. Differential efficacy of non-invasive vagus nerve stimulation for the acute treatment of episodic and chronic cluster headache: A meta-analysis. Cephalalgia. 2019 Jul;39(8):967-977. doi: 10.1177/0333102419856607. Epub 2019 Jun 10. PMID 31246132
- [Derived] Silberstein SD, Mechtler LL, Kudrow DB, Calhoun AH, McClure C, Saper JR, Liebler EJ, Rubenstein Engel E, Tepper SJ; ACT1 Study Group. Non-Invasive Vagus Nerve Stimulation for the ACute Treatment of Cluster Headache: Findings From the Randomized, Double-Blind, Sham-Controlled ACT1 Study. Headache. 2016 Sep;56(8):1317-32. doi: 10.1111/head.12896. PMID 27593728
- Available data/document: Publication — http://onlinelibrary.wiley.com/doi/10.1111/head.12896/full — Non-Invasive Vagus Nerve Stimulation for the ACute Treatment of Cluster Headache: Findings From the Randomized, Double-Blind, Sham-Controlled ACT1 Study Stephen D. Silberstein, MD; Laszlo L. Mechtler, MD; David B. Kudrow, MD; Anne H. Calhoun, MD; Candace McClure, PhD; Joel R. Saper, MD; Eric J. Liebler; Emily Rubenstein Engel, MD; Stewart J. Tepper, MD; on Behalf of the ACT1 Study Group

RESULTS

PARTICIPANT FLOW:
Groups:
- GammaCore Open Label: Non-Invasive Vagus Nerve Stimulator
  GammaCore: Treatment with active gammacore vagus nerve stimulator
Period: Phase 1 Double Blind Period
Arm/Group | Sham GammaCore Device | GammaCore Device | GammaCore Open Label
Started | 77 | 73 | 0
Completed | 58 | 42 | 0
Not Completed | 19 | 31 | 0
Period: Phase 2 Open Label
Arm/Group | Sham GammaCore Device | GammaCore Device | GammaCore Open Label
Started | 0 | 0 | 100
Completed | 0 | 0 | 74
Not Completed | 0 | 0 | 26

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham GammaCore Device | GammaCore Device | Total
Number analyzed (Participants) | 77 | 73 | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 77 | 73 | 150
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 14 | 24
  Male | 67 | 59 | 126
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 68 | 63 | 131
  Black | 7 | 5 | 12
  Asian | 1 | 4 | 5
Height [Mean (Standard Deviation); unit: inches] | 69.8 (3.84) | 69.4 (3.62) | 69.6 (3.73)
Weight [Mean (Standard Deviation); unit: pounds] | 193 (37.79) | 189.5 (40.79) | 191.3 (39.19)
CH Type [Count of Participants; unit: Participants]
  Episodic | 51 | 50 | 101
  Chronic | 26 | 23 | 49
Taking CH Prevention Medicaiton [Count of Participants; unit: Participants] | 60 | 42 | 102
Full Time Employment [Count of Participants; unit: Participants] | 47 | 45 | 92

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Repsonse to Treatment
Description: The primary outcome measurement for effectiveness is the rate of responders for the active treatment group, compared to the sham control group.
  A responder is defined as a subject who has recorded an intensity of 0 or 1 on the 5-point headache pain scale (no pain, mild, moderate, severe, very severe) at 15 minutes post-initiation of treatment of the first treated cluster headache attack of Phase 1.
Time Frame: 15 minutes post stimulation
Population: Intent to treat study population
Measure: Count of Participants; unit: Participants
Arm/Group | Sham GammaCore Device | GammaCore Device
Number analyzed (Participants) | 77 | 73
Participants
  Responder | 14 | 16
  Non-responder | 57 | 44
  Missing | 6 | 13

2. Secondary Outcome: Sustained Treatment Success at 1 Hour Post-Treatment
Description: Sustained treatment success at 1 hour post-treatment was defined as having recorded an intensity of 0 or 1 on the 5-point headache pain scale at 15 minutes and 1 hour post-initiation of treatment of the first treated cluster headache attack of Phase 1, and having refrained from use of rescue medications during the full 60 minute period
Time Frame: For 1 hour post stimulation
Measure: Count of Participants; unit: Participants
Arm/Group | Sham GammaCore Device | GammaCore Device
Number analyzed (Participants) | 77 | 73
Participants
  Yes | 9 | 16
  No | 63 | 44
  Missing | 5 | 13

3. Secondary Outcome: Average Mean Attack Intensities Experienced Per Subject
Description: Cluster headache attack intensity was reported on a 5-point scale: no pain, mild, moderate, severe, very severe, whereas no pain =1 is the best outcome and very severe=5 is the worst outcome . The average of all subjects' mean attack intensities experienced at 15 minutes post-initiation of treatment during Phase 1 for the active treatment group, compared to the sham control group. The mean 15-minute scores were calculated for the first five attacks suffered by each subject during Phase 1. For subjects with fewer than five treated attacks, the scores for those available were averaged.
Time Frame: 15 minutes post-stimulation
Population: There were 4 subjects with no data in the Sham GammaCore group and 13 subject in the GammaCore group.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sham GammaCore Device | GammaCore Device
Number analyzed (Participants) | 73 | 60
Score on a scale | 2.0 (0.9) | 2.1 (0.93)

4. Secondary Outcome: Incidence and Occurrence of Serious Adverse Events Related to Active or Sham Study Treatment and / or to Cluster Headache Events.
Description: The primary safety measure for this study is the incidence and occurrence of serious adverse events related to active or sham study treatment and / or to cluster headache events during Phase 1 of the study.
Time Frame: 4 weeks, Phase 1
Measure: Number; unit: Serious Adverse Events
Arm/Group | Sham GammaCore Device | GammaCore Device
Number analyzed (Participants) | 77 | 73
Serious Adverse Events | 0 | 0

ADVERSE EVENTS:
Groups:
- Sham GammaCore Device (Randomized Period): The Sham GammaCore device looks and operates like the Active GammaCore device, but does not deliver a therapeutic stimulation treatment.
  Sham GammaCore device: Treatment with sham stimulator
- GammaCore Device (Randomized Period); GammaCore Device (Open Label Period): Non-Invasive Vagus Nerve Stimulator
  GammaCore: Treatment with active gammacore vagus nerve stimulator
Arm/Group | Sham GammaCore Device (Randomized Period) | GammaCore Device (Randomized Period) | GammaCore Device (Open Label Period)
Serious Adverse Events (participants affected / at risk) | 0/77 | 1/73 | 5/100
Other Adverse Events (participants affected / at risk) | 21/77 | 8/73 | 20/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham GammaCore Device (Randomized Period) (N=77) | GammaCore Device (Randomized Period) (N=73) | GammaCore Device (Open Label Period) (N=100)
Mesenteric ischemia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Herniated disc (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hospitalization for cluster headache pain (Nervous system disorders) | 0 (0) | 1 (2) | 2 (2) — Not device related
Multiple left upper extremity DVT (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal aortic aneurysm (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Healthcare acquired pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Anasarca (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory failure (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Urethral trauma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Left ureteral calculus (General disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham GammaCore Device (Randomized Period) (N=77) | GammaCore Device (Randomized Period) (N=73) | GammaCore Device (Open Label Period) (N=100)
Burning Sensation during treatment (Product Issues) | 5 (5) | 0 (0) | 1 (1)
Cold/Flu (Infections and infestations) | 0 (0) | 0 (0) | 6 (7)
Dysguesia (Product Issues) | 7 (7) | 0 (0) | 2 (2)
Erythema (Product Issues) | 9 (9) | 0 (0) | 2 (2)
Myokymia (Product Issues) | 0 (0) | 8 (8) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days